CLINICAL TRIAL: NCT00523003
Title: A Controlled Trial of Protein Enrichment of Meal Replacements for Weight Reduction With Retention of Lean Body Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Zhaoping Li, Prinicpal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-06-120
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Weight Loss; Obesity
Keywords: weight loss; obesity; high protein; meal replacement
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1, (Experimental): 2.2 g protein/kg LBM/day high protein diet
  Interventions: Dietary Supplement: high protein
- 2, standard protein (Placebo Comparator): 1.1 g protein/kg LBM/day standard protein diet
  Interventions: Dietary Supplement: standard protein

INTERVENTIONS:
Dietary Supplement: high protein — 2.2 g protein/kg of LBM per day
  Arms: 1,
Dietary Supplement: standard protein — 1.1 g protein/kg LBM/day standard protein diet
  Arms: 2, standard protein

SUMMARY:
Study hypothesis: High protein diets have been shown to make people full and and help to retent of muscle mass. This study was designed to determine effects of a protein- enriched meal replacement (MR) on weight loss and muscle mass retention by comparison to an equal calorie carbohydrate-enriched MR.

Methods: Single blind, placebo-controlled, randomized outpatient weight loss trial in 100 obese men and women comparing two equal calorie meal plans.,1) 2.2 g protein/kg of LBM per day [high protein diet (HP)] or 2) 1.1 g protein/kg LBM/day standard protein diet (SP). Body weight, body composition, and lipid profiles were measured at baseline and 12 weeks.

DETAILED DESCRIPTION:
Background: While high protein diets have been shown to improve satiety and retention of lean body mass (LBM), this study was designed to determine effects of a protein- enriched meal replacement (MR) on weight loss and LBM retention by comparison to an isocaloric carbohydrate-enriched MR within customized diet plans utilizing MR to achieve high protein or standard protein intakes.

Methods: Single blind, placebo-controlled, randomized outpatient weight loss trial in 100 obese men and women comparing two isocaloric meal plans utilizing a standard MR to which was added supplementary protein or carbohydrate powder. MR were used twice daily (one meal, one snack). One additional meal was included in the meal plan designed to achieve individualized protein intakes of either 1) 2.2 g protein/kg of LBM per day [high protein diet (HP)] or 2) 1.1 g protein/kg LBM/day standard protein diet (SP). LBM was determined using bioelectrical impedance analysis (BIA). Body weight, body composition, and lipid profiles were measured at baseline and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 27 to 40 kg/m2
* in good health by history, physical examination, and basic laboratory screening (complete blood count, serum chemistries, liver panel, and lipid panel)

Exclusion Criteria:

* type 2 diabetes or glucose intolerance
* regularly drank more than one alcoholic beverage daily
* unable to provide consent

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-05 (Actual); Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 weeks

SECONDARY OUTCOMES:
Body composition, lipid panel | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — California University, Los Angeles